CLINICAL TRIAL: NCT07222826
Title: Non-invasive Intracranial Pressure Estimation by Measurement of the Occlusion Pressure of the Isolated Periorbital Vein (NICE-ICP)
Brief Title: Non-invasive Intracranial Pressure Estimation by Measurement of the Occlusion Pressure of the Isolated Periorbital Vein
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Compremium AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NICE-ICP
Record Dates: First submitted 2025-10-10; First posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Intracranial Pressure; Intracranial Pressure Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- CPMX3 Measurement (Experimental): CPMX 3 measurement
  Interventions: Device: CPMX3

INTERVENTIONS:
Device: CPMX3 — CPMX3 periorbital vein pressure measurement

SUMMARY:
Elevated intracranial pressure is a common complication of brain injury which means that the pressure within the skull rises above normal levels. The negative impact of increased intracranial pressure (ICP) on the prognosis of patients has been strongly shown in numerous studies and ICP-based treatment is associated with an important reduction of risk of death. Invasive ICP measurement methods are nowadays a standard of care in severe brain injury. The two available ways of measuring ICP require neurosurgical procedure to implant a catheter and probes within the brain and present risks and complications for the patient, such as infections and intracranial bleeding. In addition, invasive recording of ICP requires neurosurgical expertise and intensive care unit (ICU) facilities, limiting the application of ICP measurements to patients of the acute neuro-ICU (neuro-Intensive Care Unit) with acute brain damage requiring close surveillance to prevent further deterioration of neural tissue and disability. Non-invasive ICP monitoring benefits include no risk of complications seen in invasive monitoring, helping in deciding which patient needs invasive ICP monitoring, and providing ongoing long-term measurements of ICP without having to insert a new device every time. Although many non-invasive ICP measurement methods have been explored, to date, none of them have shown clinical success or usefulness. One under-explored window to ICP is the orbital vein, a small blood vessel located near your eye, which we think could provide a direct link to the intracranial pressure. The study device, called the CPMX3 system, is a non-invasive method to measure pressure in a superficial periorbital vein.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age > 18
* Equipped with an invasive ICP monitor as part of standard of care

Exclusion Criteria:

* Presence of facial and/or skull trauma that could hinder placement of the pneumatic mask or contraindicate ultrasound on the forehead
* History of recent cranial surgery or hemicraniectomy
* Active bleeding (proven or suspected)
* History or known pathological condition or injury linked to the orbital socket influencingvenous outflow (e.g. Grave disease, tumor, inflammation, trauma, glaucoma, etc.)
* History, or known vein stenosis in ophthalmic veins/cavernous sinus
* Any other condition that would interfere with measurement technique and routine clinical care according to the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety of venous pressure of the isolated periorbital vein measured with the CPMX3 System to estimate ICP, evaluated by incidence of reported adverse events | up to 7 days
Safety of venous pressure of the isolated periorbital vein measured with the CPMX3 System to estimate ICP, evaluated by incidence of reported Device Deficiencies (DDs) | Up to 7 days
Safety of venous pressure of the isolated periorbital vein measured with the CPMX3 System to estimate ICP, evaluated by incidence of reported Serious Adverse Device Effects (SADEs) | Up to 7 Days
Preliminary accuracy of venous pressure of the isolated periorbital vein measured with the CPMX3 System to estimate ICP, measured in mmHg | up to 7 days
  Preliminary accuracy will be assessed by recording paired measurements of venous occlusion pressure of the periorbital vein when isolated from its surrounding network and invasive ICP measurements from the standard of care invasive ICP monitor in mmHg

SECONDARY OUTCOMES:
Feasibility of finding and compressing the target periorbital vein as reported by the investigator using a visual analog scale 0 to 3 | up to 7 days
  As reported by investigator using a visual analog scale score from 0 to 3 (0: not able to visualize the vein, 3: perfectly able to visualize)
The tolerability of the non-invasive measurement process, evaluated via a dedicated patient questionnaire on patient comfort | up to 7 days
  Evaluated by each participant before study termination through a dedicated questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided